CLINICAL TRIAL: NCT01536899
Title: Behavioral Economic Analysis of Medical Marijuana Use in HIV+ Patients Prospective Cohort Study
Brief Title: Medical Marijuana Use in HIV+ Patients Prospective Cohort Study
Acronym: MMC-1
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor, Wayne State University
Other Study IDs: MMC-1; R01DA032678 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: HIV Positive; Marijuana Smoking
Keywords: HIV positive; Medical Marijuana
MeSH Terms: conditions — HIV Seropositivity; Marijuana Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are interested in understanding personal factors such as medical conditions and mental health, as well as social and economic factors, that influence marijuana (and other substance) use in HIV-positive patients.

Several alternative hypotheses will be evaluated in the proposed project:

1. healthier patients may self-select marijuana use;
2. marijuana use may be associated with consequences that create barriers to seeking healthcare;
3. marijuana use may have medicinal value that reduces the need for such care.

DETAILED DESCRIPTION:
The study will involve a total of 5 interviews with clinical research staff members, the total involvement will be for about 1 year.

The first interview will establish a baseline of current behaviors and health status; this will take about 3-4 hours. This interview will take place at the Tolan Park Medical Building, located at 3901 Chrysler Service Dr. The remaining 4 interviews - which will be shorter in length - will be conducted about 3, 6, 9, and 12 months after the baseline interview; each follow-up interview will take about 2 hours.The purpose of the 4 remaining interviews is to assess changes in behaviors and health status over time.

We will collect urine samples at each of the 5 interview sessions to assess health and illicit drug use.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients in the HIV clinic.
* Participants will have HIV.
* Participants will sign a single consent form.
* Participants will be marijuana users.

Exclusion Criteria:

* Participants who test negative for marijuana will be excluded.
* Volunteers who exhibit signs of drug intoxication or cognitive/mental impairment during the consent process will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive and marijuana using volunteers
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2012-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University (HIV clinic, Tolan Park Medical Buiding), Detroit, Michigan, United States

REFERENCES:
- [Derived] Woodcock EA, Greenwald MK, Chen I, Feng D, Cohn JA, Lundahl LH. HIV chronicity as a predictor of hippocampal memory deficits in daily cannabis users living with HIV. Drug Alcohol Depend Rep. 2023 Sep 13;9:100189. doi: 10.1016/j.dadr.2023.100189. eCollection 2023 Dec. PMID 37736522